CLINICAL TRIAL: NCT01610245
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Nitazoxanide and Nitazoxanide Plus Oseltamivir in the Treatment of Acute Uncomplicated Influenza
Brief Title: Safety and Efficacy Study of Nitazoxanide in the Treatment of Acute Uncomplicated Influenza
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RM08-3002
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — nitazoxanide; Oseltamivir; dolichyl-diphosphooligosaccharide - protein glycotransferase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nitazoxanide (Active Comparator): Two Nitazoxanide 300 mg tablets and one placebo capsule twice daily with food for 5 days
  Interventions: Drug: Nitazoxanide; Drug: Placebo Oral Capsule
- Oseltamivir (Active Comparator): Two placebo tablets and one Oseltamivir 75 mg capsule twice daily with food for 5 days
  Interventions: Drug: Oseltamivir; Drug: Placebo Oral Tablet
- Nitazoxanide and Oseltamivir (Active Comparator): Two nitazoxanide 300 mg tablets and one Oseltamivir 75 mg capsule twice daily with food for 5 days
  Interventions: Drug: Nitazoxanide; Drug: Oseltamivir
- Placebo (Placebo Comparator): Two placebo tablets and one placebo capsule with food twice daily for 5 days
  Interventions: Drug: Placebo Oral Tablet; Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Nitazoxanide
  Other Names: Alinia; NTZ (nitazoxanide)
  Arms: Nitazoxanide; Nitazoxanide and Oseltamivir
Drug: Oseltamivir
  Other Names: Tamiflu; OST (oseltamivir)
  Arms: Nitazoxanide and Oseltamivir; Oseltamivir
Drug: Placebo Oral Tablet
  Arms: Oseltamivir; Placebo
Drug: Placebo Oral Capsule
  Arms: Nitazoxanide; Placebo

SUMMARY:
This study is a global multicenter randomized factorial double-blind, placebo-controlled trial designed to evaluate (i) efficacy and safety of nitazoxanide 600 mg administered orally twice daily for five days compared to a placebo in the treatment of acute uncomplicated influenza and (ii) efficacy and safety of combination therapy with nitazoxanide 600 mg plus Oseltamivir 75 mg co-administered orally twice daily for five days compared to nitazoxanide monotherapy (600 mg b.i.d. for 5 days) and Oseltamivir monotherapy (75 mg b.i.d. for 5 days) in the treatment of acute uncomplicated influenza.

ELIGIBILITY:
Inclusion Criteria:

1. Age 13 to 65 years
2. Presence of clinical signs and/or symptoms consistent with acute illness compatible with influenza infection (each of the following is required):

   1. oral temperature of ≥100.4 °F or ≥38 °C (obtained in office or self-measured within 12 hours prior to screening - if self-measured, subject must also have taken an antipyretic within 4 hours prior to screening) AND
   2. at least one of the following respiratory symptoms (cough, sore throat, nasal obstruction) that is considered by the patient to be moderate or severe (greater than mild severity) AND
   3. one of the following constitutional symptoms (fatigue, headache, myalgia, feverishness) that is considered by the patient to be moderate or severe (greater than mild severity).
3. Confirmation of influenza A or B infection in the local community by one of the following means:

   1. the institution's local laboratory, or
   2. the local public health system, or
   3. the national public health system, or
   4. a laboratory of a recognized national or multinational influenza surveillance scheme.
4. Onset of illness no more than 48 hours before enrollment in the trial.

   Note: Time of onset of illness is defined as either the earlier of:
   1. the time when the temperature was first measured as elevated, OR
   2. the time when the subject experienced the presence of at least one respiratory symptom AND the presence of at least one constitutional symptom.
5. Willing and able to provide written informed consent (including assent by legal guardian if under 18 years of age) and comply with the requirements of the protocol, including completion of the patient diary.

Exclusion Criteria:

1. Severity of illness requiring or anticipated to require in-hospital care or subject defined as being at high risk of complications from influenza infection according to the Infectious Diseases Society of America (IDSA) guidelines for seasonal influenza in adults and children (Committee of Infectious Diseases (CID) 2009:48) or current Centers for Disease Control and Prevention (CDC) criteria. Current criteria for persons 13-65 years of age who are at risk of influenza complications include (list to be reviewed and updated as required prior to initiation of the study and at least monthly during the study):

   1. Persons with asthma or other chronic pulmonary diseases, such as cystic fibrosis in children or chronic obstructive pulmonary disease in adults.
   2. Persons with hemodynamically significant cardiac disease.
   3. Persons who have immunosuppressive disorders or who are receiving immunosuppressive therapy.
   4. HIV-infected persons.
   5. Persons with sickle cell anemia or other hemoglobinopathies.
   6. Persons with diseases requiring long-term aspirin therapy, such as rheumatoid arthritis or Kawasaki disease.
   7. Persons with chronic renal dysfunction.
   8. Persons with liver disorders.
   9. Persons with cancer.
   10. Persons with chronic metabolic disease, such as diabetes mellitus, inherited metabolic disorders and mitochondrial disorders.
   11. Persons with neuromuscular disorders, seizure disorders or cognitive dysfunction that may compromise the handling of respiratory secretions.
   12. Residents of any age of nursing homes or other long-term care institutions.
   13. Persons who are morbidly obese (Body Mass Index ≥40)
   14. American Indians (seemed to be at higher risk of complications last flu season)
   15. Alaskan natives (seemed to be at higher risk of complications last flu season)
2. Females of childbearing potential who are either pregnant, breast-feeding or are sexually active without the use of birth control. Female patients of child-bearing potential that are sexually active must have a negative baseline pregnancy test and must agree to continue an acceptable method of birth control for the duration of the study and for 1 month post-treatment. A double barrier method, oral birth control pills administered for at least 2 monthly cycles prior to study drug administration, an intrauterine device (IUD), or medroxyprogesterone acetate administered intramuscularly for a minimum of one month prior to study drug administration are acceptable methods of birth control for inclusion into the study. Female subjects are considered of childbearing potential unless they are postmenopausal (absence of menstrual bleeding for 1 year - or 6 months if laboratory confirmation of hormonal status), or have had a hysterectomy, bilateral tubular ligation or bilateral ovariectomy.
3. Vaccination for seasonal influenza on or after i. August 1, 2012 in the case of subjects enrolled during the 2012/2013 flu season in the United States, ii. February 1, 2013 in the case of subjects enrolled during the 2013 flu season in Australia or New Zealand, or iii. August 1, 2013 in the case of subjects enrolled during the 2013/2014 flu season in the United States, Canada, Europe, or other countries in the Northern Hemisphere, or iv. February 1, 2014 in the case of subjects enrolled during the 2014 flu season in Australia or New Zealand, or v. August 1, 2014 in the case of subjects enrolled during the 2014/2015 flu season in the United States, Canada, Europe, or other countries in the Northern Hemisphere.
4. Receipt of any dose of nitazoxanide, oseltamivir, zanamivir, amantadine, or rimantadine within 30 days prior to screening.
5. Prior treatment with any investigational drug therapy within 30 days prior to screening.
6. Subjects with active respiratory allergies or subjects expected to require anti-allergy medications during the study period for respiratory allergies.
7. Known sensitivity to Nitazoxanide or any of the excipients comprising the Nitazoxanide tablets.
8. Known sensitivity to Oseltamivir or any of the excipients comprising the Oseltamivir capsules.
9. Subjects unable to take oral medications.
10. Subject has chronic kidney or liver disease (including Hepatitis A,B or C) or known impaired hepatic and/or renal function.
11. Presence of any other pre-existing chronic infection that is undergoing or requiring medical therapy.
12. Presence of any pre-existing illness that, in the opinion of the investigator, would place the subject at an unreasonably increased risk through participation in this study.
13. Subjects who, in the judgment of the investigator, will be unlikely to comply with the requirements of this protocol.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1941 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-04-16 (Actual)

PRIMARY OUTCOMES:
Time to resolution of all clinical symptoms of influenza as reported by the subjects | Up to 28 days

SECONDARY OUTCOMES:
Time to resolution of each individual symptom of influenza | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Rossignol, M.D., Ph.D., Study Director — Romark Laboratories L.C.
Locations (154):
- United States (124):
  - Influence Study Site, Birmingham, Alabama
  - Influence Study Site, Dothan, Alabama
  - Influence Study Site, Hoover, Alabama
  - Influence Study Site, Mobile, Alabama
  - Influence Study Site, Mesa, Arizona
  - Influence Study Site, Tucson, Arizona
  - Influence Study Site, Hot Springs, Arkansas
  - Influence Study Site, Jonesboro, Arkansas
  - Influence Study Site, Anaheim, California
  - Influence Study Site, Fresno, California
  - Influence Study Site, Garden Grove, California
  - Influence Study Site, Harbor City, California
  - Influence Study Site, Huntington Beach, California
  - Influence Study Site, Lomita, California
  - Influence Study Site, Long Beach, California
  - Influence Study Site, Modesto, California
  - Influence Study Site, Norco, California
  - Influence Study Site, San Ramon, California
  - Influence Study Site, Stockton, California
  - Influence Study Site, Centennial, Colorado
  - Influence Study Site, Colorado Springs, Colorado
  - Influence Study Site, Littleton, Colorado
  - Influence Study Site, Longmont, Colorado
  - Influence Study Site, Thornton, Colorado
  - Influence Study Site, Boynton Beach, Florida
  - Influence Study Site, Coral Gables, Florida
  - Influence Study Site, Edgewater, Florida
  - Influence Study Site, Kissimmee, Florida
  - Influence Study Site, Lauderdale Lakes, Florida
  - Influence Study Site, Miami, Florida
  - Influence Study Site, Orlando, Florida
  - Influence Study Site, Pembroke Pines, Florida
  - Influence Study Site, Saint Cloud, Florida
  - Influence Study Site, West Palm Beach, Florida
  - Influence Study Site, Atlanta, Georgia
  - Influence Study Site, Canton, Georgia
  - Influence Study Site, Columbus, Georgia
  - Influence Study Site, Blackfoot, Idaho
  - Influence Study Site, Skokie, Illinois
  - Influence Study Site, Evansville, Indiana
  - Influence Study Site, Franklin, Indiana
  - Influence Study Site, Muncie, Indiana
  - Influence Study Site, Augusta, Kansas
  - Influence Study Site, Kansas City, Kansas
  - Influence Study Site, Newton, Kansas
  - Influence Study Site, Wichita, Kansas
  - Influence Study Site, Hawesville, Kentucky
  - Influence Study Site, Madisonville, Kentucky
  - Influence Study Site, Owensboro, Kentucky
  - Influence Study Site, Eunice, Louisiana
  - Influence Study Site, Lafayette, Louisiana
  - Influence Study Site, Lake Charles, Louisiana
  - Influence Study Site, Fall River, Massachusetts
  - Influence Study Site, Ann Arbor, Michigan
  - Influence Study Site, Chelsea, Michigan
  - Influence Study Site, Essexville, Michigan
  - Influence Study Site, Niles, Michigan
  - Influence Study Site, Troy, Michigan
  - Influence Study Site, Bridgeton, Missouri
  - Influence Study Site, Fremont, Nebraska
  - Influence Study Site, Las Vegas, Nevada
  - Influence Study Site, Teaneck, New Jersey
  - Influence Study Site, Albuquerque, New Mexico
  - Influence Study Site, Brooklyn, New York
  - Influence Study Site, Great Neck, New York
  - Influence Study Site, New York, New York
  - Influence Study Site, Rochester, New York
  - Influence Study Site, Westfield, New York
  - Influence Study Site, Charlotte, North Carolina
  - Influence Study Site, Hickory, North Carolina
  - Influence Study Site, Mooresville, North Carolina
  - Influence Study Site, Winston-Salem, North Carolina
  - Influence Study Site, Columbus, Ohio
  - Influence Study Site, Dayton, Ohio
  - Influence Study Site, Groveport, Ohio
  - Influence Study Site, Lyndhurst, Ohio
  - Influence Study Site, Middleburg Heights, Ohio
  - Influence Study Site, Milford, Ohio
  - Influence Study Site, Willoughby Hills, Ohio
  - Influence Study Site, Wooster, Ohio
  - Influence Study Site, Tulsa, Oklahoma
  - Influence Study Site, Ashland, Oregon
  - Influence Study Site, Gresham, Oregon
  - Influence Study Site, Altoona, Pennsylvania
  - Influence Study Site, Lansdale, Pennsylvania
  - Influence Study Site, Pittsburgh, Pennsylvania
  - Influence Study Site, Reading, Pennsylvania
  - Influence Study Site, Scottdale, Pennsylvania
  - Influence Study Site, Uniontown, Pennsylvania
  - Influence Study Site, Warwick, Rhode Island
  - Influence Study Site, Charleston, South Carolina
  - Influence Study Site, Rapid City, South Dakota
  - Influence Study Site, Bristol, Tennessee
  - Influence Study Site, Columbia, Tennessee
  - Influence Study Site, Elizabethton, Tennessee
  - Influence Study Site, Franklin, Tennessee
  - Influence Study Site, Jackson, Tennessee
  - Influence Study Site, Smyrna, Tennessee
  - Influence Study Site, Austin, Texas
  - Influence Study Site, Beaumont, Texas
  - Influence Study Site, Bryan, Texas
  - Influence Study Site, Houston, Texas
  - Influence Study Site, Irving, Texas
  - Influence Study Site, Lake Jackson, Texas
  - Influence Study Site, North Richland Hills, Texas
  - Influence Study Site, Pharr, Texas
  - Influence Study Site, Plano, Texas
  - Influence Study Site, San Antonio, Texas
  - Influence Study Site, Sugar Land, Texas
  - Influence Study Site, Waco, Texas
  - Influence Study Site, Draper, Utah
  - Influence Study Site, Magna, Utah
  - Influence Study Site, Orem, Utah
  - Influence Study Site, Salt Lake City, Utah
  - Influence Study Site, Alexandria, Virginia
  - Influence Study Site, Ashburn, Virginia
  - Influence Study Site, Charlottesville, Virginia
  - Influence Study Site, Gainesville, Virginia
  - Influence Study Site, Midlothian, Virginia
  - Influence Study Site, Norfolk, Virginia
  - Influence Study Site, Virginia Beach, Virginia
  - Influence Study Site, Port Orchard, Washington
  - Influence Study Site, Spokane, Washington
  - Influence Study Site, La Crosse, Wisconsin
- Australia (11):
  - Influence Study Site, Cardiff, New South Wales
  - Influence Study Site, Castle Hill, New South Wales
  - Influence Study Site, Darlinghurst, New South Wales
  - Influence Study Site, Westmead, Sydney, New South Wales
  - Influence Study Site, Chermside, Queensland
  - Influence Study Site, Sherwood, Queensland
  - Influence Study Site, Daw Park, South Australia
  - Influence Study Site, Clayton, Victoria
  - Influence Study Site, Fitzroy North, Victoria
  - Influence Study Site, Prahran, Victoria
  - Influence Study SIte, Nedlands, Western Australia
- Influence Study Site, Antwerp, Belgium
- Canada (11):
  - Influence Study Site, Coquitlam, British Columbia
  - Influence Study Site, Langley, British Columbia
  - Influence Study Site, Surrey, British Columbia
  - Influence Study Site, Brampton, Ontario
  - Influence Study Site, London, Ontario
  - Influence Study Site, Niagara Falls, Ontario
  - Influence Study Site, Sarnia, Ontario
  - Influence Study Site, Toronto, Ontario
  - Influence Study Site, Mirabel, Quebec
  - Influence Study Site, Montreal, Quebec
  - Influence Study Site, Pointe-Claire, Quebec
- New Zealand (7):
  - Influence Study Site, Birkenhead, Auckland
  - Influence Study Site, Grafton, Auckland
  - Influence Study Site, Remuera, Auckland
  - Influence Study Site, Rotorua, Bay of Plenty
  - Influence Study Site, Tauranga, Bay of Plenty
  - Influence Study Site, Beckenham, Christchurch
  - Influence Study Site, Christchurch Central, Christchurch